CLINICAL TRIAL: NCT04794062
Title: Myocardial Injury and Quality of Life in Patients Recovered From the Pneumonia Associated With the Novel Coronavirus Infectious Disease COVID-19
Brief Title: Myocardial Injury and Quality of Life After COVID-19
Status: Completed | Type: Observational
Sponsor: Voronezh Regional Clinical Consultative and Diagnostic Center (Network)
Collaborators: Voronezh State Medical University named after N.N. Burdenko (Other); Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Roman Khokhlov, MD, Professor, Doctor of Sciences (Dr.Sc.), Voronezh Regional Clinical Consultative and Diagnostic Center
Other Study IDs: 08092020
Record Dates: First submitted 2021-02-15; First posted 2021-03-11 (Actual); Results first posted 2024-02-15 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: COVID-19; Myocardial Injury; Myocarditis Post Infection
Keywords: COVID-9; myocardial injury; myocarditis
MeSH Terms: conditions — COVID-19; Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this observational study follow-up and dynamic observation will be conducted on the participants recovered from pneumonia caused by COVID-19. The main goal is an early diagnosis and detection of myocardial (heart) injury and quality of life in participants recovered from COVID-19 and follow-up in selected participants with present signs of myocarditis and/or myocardial fibrosis.

DETAILED DESCRIPTION:
The main goal of this observational non-interventional study is the evaluation of prevalence of myocardial injury (heart injury) of the participants recovered from the novel coronavirus infectious disease (COVID-19). Participants with signs of myocarditis (pericarditis) and/or myocardial fibrosis, and with a threat of heart failure development and other outcomes are selected into this study. In this cohort the percentage of participants having myocardial injury based on the level of high-sensitivity troponin, echocardiography (decreased Left Ventricle Ejection Fraction, abnormalities of wall motion, Right Ventricle dysfunction, increased size of heart chambers above referential values, presence of pericardial effusion), cardiac MRI with contrast enhancement (presence of edema on T2-weighted images, presence of early and late gadolinium enhancement phenomenon, local motion abnormalities, increased size of heart chambers above referential values, presence of pericardial effusion). At 6 months of the dynamic follow-up, MRI with contrast enhancement will be repeated in the participants with established myocardial injury at inclusion to assess the percentage of the participants having ongoing myocardial injury.

The secondary goal of the study is evaluation of quality of life of the patients recovered from the novel coronavirus infectious disease (COVID-19) by the means of EQ-5D and/or DASI questionnaire using the descriptive system of 5 components of quality of life related to the wellbeing, and visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of age above 18 years with diagnosed SARS-CoV-2 infection based on the PCR (polymerase chain reaction) and/or quantitative tests of IgM and IgG antibodies in serum;
* Pneumonia development confirmed by chest computed tomography;
* Negative PCR test for SARS-CoV-2 at the time of inclusion into the study;
* Stable patient state allowing outpatient follow-up;
* Signed informed consent.

Exclusion Criteria:

* Absence of convincing data confirming SARS-CoV-2 infection of a participant at the time of inclusion;
* Absence of medical records regarding previous treatment of COVID-19;
* Low compliance and unwillingness to undergo defined examinations;
* Absence of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community population of the Voronezh region in Western Russia, without need of hospitalization, sent to by the primary care physicians.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Khokhlov, MD, Principal Investigator — Voronezh Regional Clinical Consultative and Diagnostic Center
Locations (1):
- Voronezh Region Clinical, Consultative and Diagnostic Center, Voronezh, Voronezh Oblast, Russia

REFERENCES:
- [Background] Tavazzi G, Pellegrini C, Maurelli M, Belliato M, Sciutti F, Bottazzi A, Sepe PA, Resasco T, Camporotondo R, Bruno R, Baldanti F, Paolucci S, Pelenghi S, Iotti GA, Mojoli F, Arbustini E. Myocardial localization of coronavirus in COVID-19 cardiogenic shock. Eur J Heart Fail. 2020 May;22(5):911-915. doi: 10.1002/ejhf.1828. Epub 2020 Apr 11. PMID 32275347
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Rudski L, Januzzi JL, Rigolin VH, Bohula EA, Blankstein R, Patel AR, Bucciarelli-Ducci C, Vorovich E, Mukherjee M, Rao SV, Beanlands R, Villines TC, Di Carli MF; Expert Panel From the ACC Cardiovascular Imaging Leadership Council. Multimodality Imaging in Evaluation of Cardiovascular Complications in Patients With COVID-19: JACC Scientific Expert Panel. J Am Coll Cardiol. 2020 Sep 15;76(11):1345-1357. doi: 10.1016/j.jacc.2020.06.080. Epub 2020 Jul 22. PMID 32710927
- [Background] Lindner D, Fitzek A, Brauninger H, Aleshcheva G, Edler C, Meissner K, Scherschel K, Kirchhof P, Escher F, Schultheiss HP, Blankenberg S, Puschel K, Westermann D. Association of Cardiac Infection With SARS-CoV-2 in Confirmed COVID-19 Autopsy Cases. JAMA Cardiol. 2020 Nov 1;5(11):1281-1285. doi: 10.1001/jamacardio.2020.3551. PMID 32730555
- [Background] Huang L, Zhao P, Tang D, Zhu T, Han R, Zhan C, Liu W, Zeng H, Tao Q, Xia L. Cardiac Involvement in Patients Recovered From COVID-2019 Identified Using Magnetic Resonance Imaging. JACC Cardiovasc Imaging. 2020 Nov;13(11):2330-2339. doi: 10.1016/j.jcmg.2020.05.004. Epub 2020 May 12. PMID 32763118
- [Background] Puntmann VO, Carerj ML, Wieters I, Fahim M, Arendt C, Hoffmann J, Shchendrygina A, Escher F, Vasa-Nicotera M, Zeiher AM, Vehreschild M, Nagel E. Outcomes of Cardiovascular Magnetic Resonance Imaging in Patients Recently Recovered From Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Nov 1;5(11):1265-1273. doi: 10.1001/jamacardio.2020.3557. PMID 32730619
- [Background] Hendren NS, Drazner MH, Bozkurt B, Cooper LT Jr. Description and Proposed Management of the Acute COVID-19 Cardiovascular Syndrome. Circulation. 2020 Jun 9;141(23):1903-1914. doi: 10.1161/CIRCULATIONAHA.120.047349. Epub 2020 Apr 16. PMID 32297796
- [Background] Medical rehabilitation during the novel coronavirus 19 disease (COVID-19). Physical and rehabilitation medicine, medical rehabilitation. 2020;2(2):140-189. DOI: https://doi.org/10.36425/rehab34231
- [Background] Temporary methodical recommendation "Prophylaxis, diagnosis, and treatment of the novel coronavirus 19 (COVID-19)", 9th Edition released on 10/26/2020
- [Background] Schultz JC, Hilliard AA, Cooper LT Jr, Rihal CS. Diagnosis and treatment of viral myocarditis. Mayo Clin Proc. 2009 Nov;84(11):1001-9. doi: 10.1016/S0025-6196(11)60670-8. PMID 19880690
- [Background] Friedrich MG, Sechtem U, Schulz-Menger J, Holmvang G, Alakija P, Cooper LT, White JA, Abdel-Aty H, Gutberlet M, Prasad S, Aletras A, Laissy JP, Paterson I, Filipchuk NG, Kumar A, Pauschinger M, Liu P; International Consensus Group on Cardiovascular Magnetic Resonance in Myocarditis. Cardiovascular magnetic resonance in myocarditis: A JACC White Paper. J Am Coll Cardiol. 2009 Apr 28;53(17):1475-87. doi: 10.1016/j.jacc.2009.02.007. PMID 19389557
- [Background] Ferreira VM, Schulz-Menger J, Holmvang G, Kramer CM, Carbone I, Sechtem U, Kindermann I, Gutberlet M, Cooper LT, Liu P, Friedrich MG. Cardiovascular Magnetic Resonance in Nonischemic Myocardial Inflammation: Expert Recommendations. J Am Coll Cardiol. 2018 Dec 18;72(24):3158-3176. doi: 10.1016/j.jacc.2018.09.072. PMID 30545455
- [Background] Caforio AL, Pankuweit S, Arbustini E, Basso C, Gimeno-Blanes J, Felix SB, Fu M, Helio T, Heymans S, Jahns R, Klingel K, Linhart A, Maisch B, McKenna W, Mogensen J, Pinto YM, Ristic A, Schultheiss HP, Seggewiss H, Tavazzi L, Thiene G, Yilmaz A, Charron P, Elliott PM; European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Current state of knowledge on aetiology, diagnosis, management, and therapy of myocarditis: a position statement of the European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2013 Sep;34(33):2636-48, 2648a-2648d. doi: 10.1093/eurheartj/eht210. Epub 2013 Jul 3. PMID 23824828
- [Background] Comparative investigation of informative yield of non-invasive diagnostics methods of inflammatory diseases of myocardium. Russian cardiology journal 2018, (154): 53-59. http://dx.doi.org/10.15829/1560-4071-2018-2-53-59
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Guidelines for the management of myocarditis. Eurasian cardiology journal 2015;3:5-17
- [Background] Giustino G, Croft LB, Stefanini GG, Bragato R, Silbiger JJ, Vicenzi M, Danilov T, Kukar N, Shaban N, Kini A, Camaj A, Bienstock SW, Rashed ER, Rahman K, Oates CP, Buckley S, Elbaum LS, Arkonac D, Fiter R, Singh R, Li E, Razuk V, Robinson SE, Miller M, Bier B, Donghi V, Pisaniello M, Mantovani R, Pinto G, Rota I, Baggio S, Chiarito M, Fazzari F, Cusmano I, Curzi M, Ro R, Malick W, Kamran M, Kohli-Seth R, Bassily-Marcus AM, Neibart E, Serrao G, Perk G, Mancini D, Reddy VY, Pinney SP, Dangas G, Blasi F, Sharma SK, Mehran R, Condorelli G, Stone GW, Fuster V, Lerakis S, Goldman ME. Characterization of Myocardial Injury in Patients With COVID-19. J Am Coll Cardiol. 2020 Nov 3;76(18):2043-2055. doi: 10.1016/j.jacc.2020.08.069. PMID 33121710
- [Background] Life quality of the Russian population by the data from ESSE-RF study. Cardiovascular Therapy and Prevention, 2016; 15(5): 84-90 http://dx.doi.org/10.15829/1728-8800-2016-5-84-90
- [Background] Health-related quality of life population indicators using EQ-5D questionnaire. Zdravookhranenie Rossiiskoi Federatsii (Health Care of the Russian Federation, Russian journal). 2018; 62(6): 295-303. (In Russ.) DOI: http://dx.doi.org/10.18821/0044-197Х-2018-62-6-295-303
- [Background] Kotecha T, Knight DS, Razvi Y, Kumar K, Vimalesvaran K, Thornton G, Patel R, Chacko L, Brown JT, Coyle C, Leith D, Shetye A, Ariff B, Bell R, Captur G, Coleman M, Goldring J, Gopalan D, Heightman M, Hillman T, Howard L, Jacobs M, Jeetley PS, Kanagaratnam P, Kon OM, Lamb LE, Manisty CH, Mathurdas P, Mayet J, Negus R, Patel N, Pierce I, Russell G, Wolff A, Xue H, Kellman P, Moon JC, Treibel TA, Cole GD, Fontana M. Patterns of myocardial injury in recovered troponin-positive COVID-19 patients assessed by cardiovascular magnetic resonance. Eur Heart J. 2021 May 14;42(19):1866-1878. doi: 10.1093/eurheartj/ehab075. PMID 33596594
- [Background] Petersen SE, Khanji MY, Plein S, Lancellotti P, Bucciarelli-Ducci C. European Association of Cardiovascular Imaging expert consensus paper: a comprehensive review of cardiovascular magnetic resonance normal values of cardiac chamber size and aortic root in adults and recommendations for grading severity. Eur Heart J Cardiovasc Imaging. 2019 Dec 1;20(12):1321-1331. doi: 10.1093/ehjci/jez232. PMID 31544926
- [Background] Douglas PS, Carabello BA, Lang RM, Lopez L, Pellikka PA, Picard MH, Thomas JD, Varghese P, Wang TY, Weissman NJ, Wilgus R. 2019 ACC/AHA/ASE Key Data Elements and Definitions for Transthoracic Echocardiography: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Data Standards (Writing Committee to Develop Cardiovascular Endpoints Data Standards) and the American Society of Echocardiography. J Am Coll Cardiol. 2019 Jul 23;74(3):403-469. doi: 10.1016/j.jacc.2019.02.027. Epub 2019 Jun 24. No abstract available. PMID 31248701
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Background] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Popescu BA, Waggoner AD. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2016 Apr;29(4):277-314. doi: 10.1016/j.echo.2016.01.011. No abstract available. PMID 27037982
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] Klein AL, Abbara S, Agler DA, Appleton CP, Asher CR, Hoit B, Hung J, Garcia MJ, Kronzon I, Oh JK, Rodriguez ER, Schaff HV, Schoenhagen P, Tan CD, White RD. American Society of Echocardiography clinical recommendations for multimodality cardiovascular imaging of patients with pericardial disease: endorsed by the Society for Cardiovascular Magnetic Resonance and Society of Cardiovascular Computed Tomography. J Am Soc Echocardiogr. 2013 Sep;26(9):965-1012.e15. doi: 10.1016/j.echo.2013.06.023. No abstract available. PMID 23998693
- [Background] Devlin NJ, Brooks R. EQ-5D and the EuroQol Group: Past, Present and Future. Appl Health Econ Health Policy. 2017 Apr;15(2):127-137. doi: 10.1007/s40258-017-0310-5. PMID 28194657
- [Background] Alexandrova E.A., Herry J. Populational indicators of quality of life related to the health according to EQ-5D questionnaire. Healthcare of the Russian Federation. 2018; 62(6): 295-303. DOI: http://dx.doi.org/10.18821/0044-197Х-2018-62-6-295-303.
- [Background] Hlatky MA, Boineau RE, Higginbotham MB, Lee KL, Mark DB, Califf RM, Cobb FR, Pryor DB. A brief self-administered questionnaire to determine functional capacity (the Duke Activity Status Index). Am J Cardiol. 1989 Sep 15;64(10):651-4. doi: 10.1016/0002-9149(89)90496-7. PMID 2782256
- See also: Manuscript published at a journal Kardiologia — https://lib.ossn.ru/jour/article/view/2268

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Recovered From COVID-19: Patients who recovered from COVID-19 and had a history of a positive polymerase chain reaction (PCR) test for SARS-CoV-2 (based on the data of the regional medical database).
Period: Overall Study
Arm/Group | Patients Recovered From COVID-19
Started | 119
Completed | 106
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Patients Recovered From COVID-19
Number analyzed (Participants) | 106
Age, Continuous [Median (Full Range); unit: years] | 57.5 [49 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 106
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Russia | 106

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients (%) Recovered From COVID-19 With a Decrease in the Global Contractility of the Left and Right Ventricles.
Description: Decrease of the left ventricle ejection fraction below 57% in men and women or decrease of the right ventricle ejection fraction below 52% in men and 51% in women.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Patients Recovered From COVID-19: Patients who recovered from COVID-19 and had a history of a positive polymerase chain reaction (PCR) test for SARS-CoV-2 (based on the data of the regional medical database).
  The main inclusion criteria were:
  1) age above 18 years and a confirmation of COVID-19 according to regional PCR database (quantitative determination of the titer of IgG/M antibodies in some cases); 2) negative result of a control PCR at the time of inclusion to the study; 3) stable medical condition of a participant, which allows examination on an outpatient basis; 4) signed informed consent.
Arm/Group | Patients Recovered From COVID-19
Number analyzed (Participants) | 106
Participants
  Decreased function of left ventricle | 19
  Decreased function of right ventricle | 39
  No decrease in left or right ventricle function | 48

2. Primary Outcome: Proportion of Patients (%) Recovered From COVID-19 With Signs of Pericardial Effusion.
Description: Presence of pericardial effusion, i.e., presence of free echocardiographic spaces between the pericardial layers during diastole with pericardial layer thickness more than 4mm.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Recovered From COVID-19
Number analyzed (Participants) | 106
Participants
  Pericardial effusion | 27
  No pericardial effusion | 79

3. Primary Outcome: Proportion of Patients (%) Recovered From COVID-19 With Signs of Early and Late Gadolinium Enhancement of Myocardium.
Description: Presence of early and late gadolinium enhancement of myocardium on cardiac MRI.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Recovered From COVID-19
Number analyzed (Participants) | 106
Participants
  Presence of early and late gadolinium enhancement of myocardium. | 28
  No early and late gadolinium enhancement of myocardium. | 78

4. Post Hoc Outcome: Evaluation of Quality of Life of the Patients Recovered From the COVID-19 by the Duke Activity Status Index.
Description: The Duke Activity Status Index is an assessment tool used to evaluate the functional capacity of patients with cardiovascular disease. Positive responses are summed up to get a total score, which ranges from 0 to 58.2. Higher scores would indicate a higher functional capacity.
Time Frame: At the time of enrollment, but analysis of quality of life criteria was additionally decided to be performed as a separate sub-study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Patients Recovered From COVID-19: Patients who recovered from COVID-19 and had a history of a positive polymerase chain reaction (PCR) test for SARS-CoV-2 (based on the data of the regional medical database).
  Patients filled a Duke Activity Status Index (DASI) score questionnaire at the time of enrollment.
Arm/Group | Patients Recovered From COVID-19
Number analyzed (Participants) | 100
units on a scale | 31.8 (12.3)

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 year
Arm/Group | Patients Recovered From COVID-19
All-Cause Mortality (participants affected / at risk) | 0/106
Serious Adverse Events (participants affected / at risk) | 0/106
Other Adverse Events (participants affected / at risk) | 0/106

LIMITATIONS AND CAVEATS:
This was a single-center, non-comparative study. Despite simple inclusion criteria for the patients recovered from COVID-19, the results of the study do not completely exclude bias. This is a cross-sectional study, which makes it impractical to describe the natural evolution of the changes found after COVID-19. The relatively small sample size makes it more difficult to compare subgroups and may prevent the identification of factors associated with heart injury and other patterns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT04794062/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT04794062/ICF_001.pdf